CLINICAL TRIAL: NCT02042898
Title: An International, Multi-centre, Randomized Controlled Trial to Assess Transfusion Thresholds in Patients Undergoing Cardiac Surgery
Brief Title: Transfusion Requirements in Cardiac Surgery III
Acronym: TRICS-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TRICSIII; 301852 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2014-01-17; First posted 2014-01-23 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Disorder; Heart, Functional, Postoperative, Cardiac Surgery
Keywords: Cardiac Surgery; Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive transfusion strategy (Active Comparator): Restrictive transfusion strategy: patients will receive a red cell transfusion if their hemoglobin is <75 g/L (<7.5 g/dL;<4.7mmol/L) intraoperatively and/or postoperatively
  Interventions: Other: Restrictive Transfusion Strategy
- Liberal transfusion strategy (Active Comparator): Liberal transfusion strategy: patients will receive a red cell transfusion if their hemoglobin concentration is <95 g/L (<9.5 g/dL<5.9mmol/L) intraoperatively, or postoperatively in the intensive care unit; and/or <85 g/L (< 8.5 g/dL;<5.3mmol/L) on the ward.
  Interventions: Other: Liberal transfusion strategy

INTERVENTIONS:
Other: Restrictive Transfusion Strategy
  Arms: Restrictive transfusion strategy
Other: Liberal transfusion strategy
  Arms: Liberal transfusion strategy

SUMMARY:
TRICS-III is an international, multi-centre, open-label randomized controlled trial of two commonly used transfusion strategies in high risk patients having cardiac surgery using a non-inferiority trial design.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Planned cardiac surgery using cardiopulmonary bypass
* Informed consent obtained
* Preoperative European System for Cardiac Operative Risk Evaluation (EuroSCORE I) of 6 or more

Exclusion Criteria:

* Patients who are unable to receive or who refuse blood products
* Patients who are involved in a preoperative autologous pre-donation program
* Patients who are having a heart transplant or having surgery solely for an insertion of a ventricular assist device
* Pregnancy or lactation (a negative pregnancy test must be obtained prior to randomization for women of childbearing potential.)
* Patients who are unable to receive or who refuse blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5028 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Composite score of any one of the following: (1) all-cause mortality; (2) myocardial infarction; (3) new renal failure requiring dialysis; or (4) new focal neurological deficit | Up to hospital discharge or postoperative day 28 (whichever occurs first)
  Composite score of any one of the following events occurring during the index hospitalization (from the start of surgery until hospital discharge or postoperative day 28, whichever comes first): (1) all-cause mortality; (2) myocardial infarction; (3) new renal failure requiring dialysis; or (4) new focal neurological deficit

SECONDARY OUTCOMES:
Incidence of in-hospital all-cause mortality | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of in-hospital myocardial infarction | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of in-hospital new renal failure requiring dialysis | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of in-hospital new focal neurological deficit | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Length of stay in the ICU and hospital | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Prolonged low output state defined as the need for two or more inotropes for 24 hours or more, intra-aortic balloon pump postoperatively or ventricular assist device | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Duration of mechanical ventilation | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of infection | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Acute kidney injury (defined by Kidney Disease Improving Global Outcomes criteria) | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of gut infarction | Up to hospital discharge or postoperative day 28 (whichever occurs first)
The proportion of patients transfused and the number of blood products and hemostatic products utilized (e.g. red cells, plasma, platelets, cryoprecipitate, factor VII) (index hospitalization) | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Death | 6 months
New onset dialysis (since incident surgery) status | 6 months
Stroke | 6 months
Coronary revascularization | 6 months
Myocardial infarction | 6 months
Health Care Utilization | 6 months
Renal function, based on changes in postoperative serum creatinine | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of Seizures | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of Encephalopathy | Up to hospital discharge or postoperative day 28 (whichever occurs first)
Incidence of Delirium | Up to hospital discharge or postoperative day 28 (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto; Nadine Shehata, MD, Principal Investigator — MOUNT SINAI HOSPITAL; Richard Whitlock, MD, Principal Investigator — McMaster University; Dean Fergusson, MD, Principal Investigator — Ottawa Hospital Research Institute; Kevin Thorpe, MSc, Principal Investigator — University of Toronto
Locations (74):
- United States (8):
  - San Francisco VA Medical Center, San Francisco, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Maine Medical Center, Portland, Maine
  - Montefiore Medical Center, The Bronx, New York
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas
- Australia (12):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Cabrini Health, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Barwon Health (University Hospital Geelong), Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Hospital Unimed Rio (National Institute of Cardiology), Rio de Janeiro, Brazil
- Canada (22):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Kelowna General Hospital, Kelowna, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - St Boniface Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Health Sciences Centre (Memorial University), St. John's, Newfoundland and Labrador
  - QEII Health Science Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Center, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network Toronto General Hospital, Toronto, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Chemin Sainte-Foy, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - SMBD Jewish General Hospital, Montreal, Quebec
  - Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- China (2):
  - Shanghai Yodak Cardio-Thoracic Hospital, Shanghai
  - Renji Hospital, Shanghai
- Colombia (5):
  - Instituto del Corazón de Bucaramanga, Bucaramanga, Santander Department
  - Clinica de Marly, Bogotá
  - Fundacion Cardioinfantil Instituto de Cardiologia, Bogotá
  - Fundación Clínica Shaio, Bogotá
  - Hospital De San Jose, Bogotá
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Tanta University Hospital, Tanta, Egypt
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Hospital Giessen, Giessen
- University of Thessaly, Volos, Greece
- India (2):
  - Narayana Health, Bangalore, Karnataka
  - SAL Hospital, Gujarat
- Israel (2):
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Centre, Tel Aviv
- Institut Jantung Negara, Kuala Lampur, Malaysia
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Wellington Hospital, Wellington
- Emergency Institute for Cardiovascular Diseases, Târgu Mureş, Romania
- National Heart Centre Singapore, Singapore, Singapore
- University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Ramón y Cajal, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Instituto de Investigación Sanitaria Hospital Univ. & Politc. La Fe de Valencia, Valencia
- Switzerland (2):
  - University Hospital Basel, Basel
  - University Hospital Bern (Inselspital), Bern

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Mistry N, Hare GMT, Shehata N, Kramer RS, Fawzy HF, Baker RA, Carmona P, Saczkowski R, Filipescu D, Alphonsus CS, Rochon A, Gregory AJ, Khanykin B, Leff JD, Mateo E, Karangelis D, Tellez JC, Saha T, Ko DT, Wijeysundera DN, Verma S, Mazer CD. Methemoglobin as a marker of acute anemic stress in cardiac surgery. iScience. 2023 Jul 20;26(8):107429. doi: 10.1016/j.isci.2023.107429. eCollection 2023 Aug 18. PMID 37575193
- [Derived] Sankar A, Rotstein AJ, Teja B, Carrier FM, Belley-Cote EP, Bolliger D, Saha T, Carmona P, Sander M, Shehata N, Thorpe KE, Mazer CD. Prolonged mechanical ventilation after cardiac surgery: substudy of the Transfusion Requirements in Cardiac Surgery III trial. Can J Anaesth. 2022 Dec;69(12):1493-1506. doi: 10.1007/s12630-022-02319-9. Epub 2022 Sep 19. PMID 36123418
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Mazer CD, Whitlock RP, Fergusson DA, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, Carrier FM, McGuinness S, Young PJ, Byrne K, Villar JC, Royse A, Grocott HP, Seeberger MD, Mehta C, Lellouche F, Hare GMT, Painter TW, Fremes S, Syed S, Bagshaw SM, Hwang NC, Royse C, Hall J, Dai D, Mistry N, Thorpe K, Verma S, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Six-Month Outcomes after Restrictive or Liberal Transfusion for Cardiac Surgery. N Engl J Med. 2018 Sep 27;379(13):1224-1233. doi: 10.1056/NEJMoa1808561. Epub 2018 Aug 26. PMID 30146969
- [Derived] Garg AX, Shehata N, McGuinness S, Whitlock R, Fergusson D, Wald R, Parikh C, Bagshaw SM, Khanykin B, Gregory A, Syed S, Hare GMT, Cuerden MS, Thorpe KE, Hall J, Verma S, Roshanov PS, Sontrop JM, Mazer CD. Risk of Acute Kidney Injury in Patients Randomized to a Restrictive Versus Liberal Approach to Red Blood Cell Transfusion in Cardiac Surgery: A Substudy Protocol of the Transfusion Requirements in Cardiac Surgery III Noninferiority Trial. Can J Kidney Health Dis. 2018 Jan 3;5:2054358117749532. doi: 10.1177/2054358117749532. eCollection 2018. PMID 29326843
- [Derived] Shehata N, Whitlock R, Fergusson DA, Thorpe KE, MacAdams C, Grocott HP, Rubens F, Fremes S, Lellouche F, Bagshaw S, Royse A, Rosseel PM, Hare G, Medicis E, Hudson C, Belley-Cote E, Bainbridge D, Kent B, Shaw A, Byrne K, Syed S, Royse CF, McGuiness S, Hall J, Mazer CD. Transfusion Requirements in Cardiac Surgery III (TRICS III): Study Design of a Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):121-129. doi: 10.1053/j.jvca.2017.10.036. Epub 2017 Nov 3. PMID 29273477
- [Derived] Mazer CD, Whitlock RP, Fergusson DA, Hall J, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, McGuinness S, Royse A, Carrier FM, Young PJ, Villar JC, Grocott HP, Seeberger MD, Fremes S, Lellouche F, Syed S, Byrne K, Bagshaw SM, Hwang NC, Mehta C, Painter TW, Royse C, Verma S, Hare GMT, Cohen A, Thorpe KE, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Restrictive or Liberal Red-Cell Transfusion for Cardiac Surgery. N Engl J Med. 2017 Nov 30;377(22):2133-2144. doi: 10.1056/NEJMoa1711818. Epub 2017 Nov 12. PMID 29130845